CLINICAL TRIAL: NCT02215473
Title: Influence of Pre-procedural Oral Rinse in the Induced Bacteremia by Periodontal Instrumentation: a Randomized Clinical Trial
Brief Title: Bacteremia in Periodontal Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Taubate (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BPP
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Gingivitis; Periodontitis
Keywords: gingivitis; periodontitis; mouth rinse; bacteremia
MeSH Terms: conditions — Gingivitis; Periodontitis; Bacteremia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- gingivitis mouth rinse (Experimental)
  Interventions: Drug: Chlorhexidine gluconate mouth rinse; Procedure: Periodontal instrumentation
- periodontitis mouth rinse (Experimental)
  Interventions: Drug: Chlorhexidine gluconate mouth rinse; Procedure: Periodontal instrumentation
- gingivitis no mouth rinse (Active Comparator)
  Interventions: Procedure: Periodontal instrumentation
- periodontitis no mouth rinse (Active Comparator)
  Interventions: Procedure: Periodontal instrumentation

INTERVENTIONS:
Drug: Chlorhexidine gluconate mouth rinse — Before local oral anesthesia and periodontal instrumentation individuals performed a single oral rinse (15mL of 0.12% chlorhexidine gluconate for 30 seconds). Debridement procedures were carried out with manual Gracey and McCall curettes and Hirschfield files.
  Arms: gingivitis mouth rinse; periodontitis mouth rinse
Procedure: Periodontal instrumentation — Individuals only received local oral anesthesia before periodontal instrumentation. Debridement procedures were carried out with manual Gracey and McCall curettes and Hirschfield files.

SUMMARY:
Bacteremia represents the presence of live germs in the blood stream. Patients with gum disease show damaged tissues and seem to be more susceptible to bacteremia. In fact, daily activities such as mastication can induce bacteremia in these patients. Dental procedures related to bleeding also induce bacteremia. However, there are many questions that should be clarified. Among them, clinical strategies that are able to reduce the levels of germs in blood should be determined. This desirable effect could be particularly important for some patients, for example, for those at higher risk for endocarditis. Therefore, this study tested if 0.12% chlorhexidine solution used as a single mouth rinse before dental instrumentation could reduce the levels of bacteria in the blood. In addition, the occurrence and magnitude of bacteremia in patients with gum disease were investigated by two different laboratorial techniques. After receiving verbal and written explanations and after signed the informed consent form, 80 systemically healthy volunteers diagnosed with gum disease having dental plaque and tartar were randomly allocated in one the following groups: a) mouth-rinse use and dental instrumentation and b) dental instrumentation with no mouth rinse. In a preliminary visit volunteers underwent a complete periodontal examination which included clinical measurements (inflammatory and debris accumulation indicators), microbial (tongue and dental plaque samples collected with paper points), saliva (to determine volume and biological indicators) and gingival crevicular fluid sampling (to monitor gingival inflammation profile). In the next visit, dental instrumentation was performed under local anesthesia, after the mouth rinse single use in the most diseased periodontal teeth/quadrant. Blood samples were collected before any dental procedure, 2 and 6 minutes after dental instrumentation. Oral hygiene instructions and periodontal treatment were performed in additional visits according to individual needs. Finally, the relation between bacteremia and several indicators of periodontal status was investigated.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate plaque related gingivitis (gingivitis group)
* mild to moderate periodontitis (periodontitis group)
* at least 20 natural teeth
* with no recognized systemic risk related to bacteremia
* no need for antibiotic prophylaxis before dental procedures

Exclusion Criteria:

* systemic diseases or other conditions that could influence the periodontal status;
* alcohol or other drugs abuse;
* orthodontic devices;
* extended prosthetic fixed devices, removable partial dentures or overhanging restorations;
* pregnancy or breast-feeding;
* history of sensitivity or suspected allergies following the use of chlorhexidine;
* antibiotics and/or anti-inflammatory drug use in the three months prior to the beginning of the study;
* regular use of chemotherapeutic antiplaque/antigingivitis products;
* any furcation lesions;
* periodontal treatment performed within six months prior to study initiation;
* unwillingness to return for follow-up.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes on viable bacterial levels in blood | 2 and 6 minutes
  To check a possible antimicrobial effect after a single mouth rinse use, the levels of viable anaerobic and aerobic bacterial cels were compared between 0 and 2 minutes, 0 and 6 minutes and between 2 and 6 minutes. Blood samples were collected and spread out onto agar plates to determine total levels of aerobic and anaerobic bacteria. Bacterial levels at 2 and 6 minutes were compared between volunteers who performed the pre-procedural rinse and who not.

SECONDARY OUTCOMES:
Changes on levels of bacterial DNA in blood | 2 and 6 months
  To check a possible antimicrobial effect after a single mouth rinse use, the levels of bacterial DNA in blood samples were compared between 0 and 2 minutes, 0 and 6 minutes and between 2 and 6 minutes. Blood samples were collected and analyzed by real time PCR (polymerase chain reaction) to determine total bacterial load and levels of target periodontal pathogens. Bacterial levels at 2 and 6 minutes were compared between volunteers who performed the pre-procedural rinse and who not.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Cortelli, PhD, Principal Investigator — University of Taubate
Locations (1):
- Nucleus of periodontal research of University of Taubate, Taubaté, São Paulo, Brazil